CLINICAL TRIAL: NCT02291133
Title: Treatment of Primary Liver Tumors With Electrochemotherapy (ECT)
Acronym: ECT-HCC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Masa Bosnjak (Other)
Collaborators: Institute of Oncology Ljubljana (Other); University of Ljubljana (Other)
Responsible Party: Sponsor-Investigator, Masa Bosnjak, PhD, MPharm, University Medical Centre Ljubljana
Organization: University Medical Centre Ljubljana (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21K/02/14
Record Dates: First submitted 2014-11-06; First posted 2014-11-14 (Estimated); Results first posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Liver Cancer
Keywords: Primary liver tumors; Bleomycin; Electrochemotherapy
MeSH Terms: conditions — Liver Neoplasms | interventions — Electrochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Electrochemotherapy treatment (Experimental)
  Interventions: Procedure: Electrochemotherapy; Device: Cliniporator Vitae®; Drug: Bleomycin PHC 15 e. (United States Pharmacopeia - USP)

INTERVENTIONS:
Procedure: Electrochemotherapy — Exploration, anesthesia, adhesiolysis, mobilization of liver, intra-operative US or CT, bleomycin administration, electroporation
Device: Cliniporator Vitae® — Positioning of electrodes, 8-28 min after administration of bleomycin application of electric pulses (8 pulses, duration 100 microseconds, frequency 8 Hz with amplitude adequate to cover the whole treated lesion with electric field necessary for reversible plasma membrane permeabilization), removal of electrodes.
  The maximum duration of procedure is 90 minutes, after liver mobilization.
Drug: Bleomycin PHC 15 e. (United States Pharmacopeia - USP) — Intravenous in bolus administration of bleomycin (15 mg/m2)

SUMMARY:
The aim of the study is to evaluate toxicity and effectiveness of electrochemotherapy with bleomycin in treatment of primary liver tumors in clinical study phase I and II.

The study will include 10 patients in phase I clinical study and additional 15 patients in phase II clinical study (or in the extension of the clinical study), which will fulfill inclusion criteria.

Treatment effectiveness will be evaluated by DCE-US or CT perfusion, to detect early events in tumor perfusion after ECT compared to tumor perfusion before ECT. Long term effectiveness of the treatment will be evaluated by modified RECIST criteria, which will take into account difference in size and density, determined from images obtained by CT perfusion of the treated tumor nodules before and after ECT. Tumor volume will be calculated by following formula , where a will be shorter and b longer tumor diameter.

The secondary objectives of the trial are to quantify the impact of the treatment on the patient's quality of life, tolerance to the therapy and suitability for larger study to be conducted.

DETAILED DESCRIPTION:
The study will be conducted on patients with primary liver tumors. 10 patients will be included in phase I clinical study and additional 15 patients in phase II clinical study (or in the extension of the clinical study).

Depending on the position of tumors, appropriate electrodes will be selected; hexagonal needle electrodes with fixed geometry for tumors not larger than 3 cm in diameter, where lower edge of the tumor is located up to 3 cm below the liver capsule or longer single needle electrodes. Individual electrodes, positioned according to the prepared treatment plan will be used for tumors up to 7 cm in diameter, or located near vena cava or large hepatic or portal veins.

Electrochemotherapy will be performed within 8-28 min after intravenous in bolus administration of bleomycin (15 mg/m2).

Triggering of electric pulses will be synchronized with ECG signals, through the ECG triggering device AccuSync to avoid delivery of pulses in vulnerable period of the heart.

All patients will be treated after the procedure has been thoroughly described to them, and have signed informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary liver tumors; hepatocellular carcinoma, intrahepatic cholangiocarcinoma and other primary tumors not larger than 7 cm that are positioned in unresectable liver area, near blood vessels in operable patients.
2. Patients with the progression of the disease (confirmed by radiological imaging) after treatment with TACE, RFA or percutaneous alcohol ablation, which are not suitable for potentially curative treatment, but with relatively good "performance status" and Child-Pugh score < 8.

   Patients from group 1. and 2. are patients, in whom standard treatment procedures are not eligible, so ECT will be the only therapeutic option. In patients with multiple liver tumors, unresectable tumors which are also unsuitable for RAF will be treated by ECT, whereas other tumors will be resected or treated by RAF.
3. Patients with tumors smaller tumors, not suitable for liver transplantation, but also unsuitable for RFA treatment or percutaneous alcohol ablation because of the position of the tumor. Electrochemotherapy will be as bridge therapy, till liver transplantation.
4. Patients with tumors> 4 cm in diameter, in difficult to reach locations, and patients unsuitable for treatment with other treatment options.

   Patients from group 3. and 4. are patients, potentially curable with standard treatment. Electrochemotherapy in these patients will not affect the standard of care of these patients, recommended in guidelines for HCC.
5. Electrochemotherapy is offered to the patients also when they refuse standard treatments.
6. Histologically confirmed primary liver cancer and/or based on radiological imaging laboratory tests confirmed primary liver cancer by multidisciplinary team for liver tumors.
7. Age more than 18.
8. Life expectancy more than 3 month.
9. Performance status Karnofsky ≥ 70 or (World Health Organization) WHO < or 2.
10. Treatment free interval 2-5 weeks, depending on the drugs used.
11. Patient must be mentally capable of understanding the information given.
12. Patient must give informed consent.
13. Patient must be discussed at the multidisciplinary team for liver tumors before entering the trial.

Exclusion Criteria:

1. Secondary primary tumor, except surgically treated noninvasive cancer of cervix, or surgically or irradiated basal cell carcinoma
2. Visceral, bone or diffuse metastases.
3. Life-threatening infection and/or heart failure and/or liver failure and/or other severe systemic pathologies.
4. Clinically significant ascites.
5. Significant reduction in respiratory function.
6. Age less than 18 years.
7. Coagulation disturbances (those who do not respond on standard treatment with vitamin-K or fresh frozen plasma).
8. Cumulative dose of 250 mg/m2 bleomycin received.
9. Allergic reaction to bleomycin.
10. Impaired kidney function (creatinin > 150 µmol/l).
11. Patients with epilepsy.
12. Patients with arrhythmias.
13. Patients with heart failure or pace maker.
14. Pregnancy.
15. Patient incapable of understanding the aim of the study or disagree with the entering into the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-06; Primary Completion 2019-09 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mihajlo Djokic, MD, Principal Investigator — University Medical Centre Ljubljana, Ljubljana, Slovenia; Blaz Trotovsek, MD, PhD, Principal Investigator — University Medical Centre Ljubljana, Ljubljana, Slovenia; Gregor Sersa, PhD, Study Director — Institute of Oncology Ljubljana, Slovenia; Borut Stabuc, MD, PhD, Study Director — University Medical Centre Ljubljana, Ljubljana, Slovenia; Dragoje Stanisavljevic, MD, Study Chair — University Medical Centre Ljubljana, Ljubljana, Slovenia; Valentin Sojar, MD, PhD, Study Chair — University Medical Centre Ljubljana, Ljubljana, Slovenia
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia, Ljubljana, Slovenia

REFERENCES:
- [Background] Edhemovic I, Brecelj E, Gasljevic G, Marolt Music M, Gorjup V, Mali B, Jarm T, Kos B, Pavliha D, Grcar Kuzmanov B, Cemazar M, Snoj M, Miklavcic D, Gadzijev EM, Sersa G. Intraoperative electrochemotherapy of colorectal liver metastases. J Surg Oncol. 2014 Sep;110(3):320-7. doi: 10.1002/jso.23625. Epub 2014 Apr 30. PMID 24782355

RESULTS

PARTICIPANT FLOW:
Groups:
- Electrochemotherapy Treatment: Electrochemotherapy: Exploration, anesthesia, adhesiolysis, mobilization of liver, intra-operative US or CT, bleomycin administration, electroporation
  Cliniporator Vitae®: Positioning of electrodes, 8-28 min after administration of bleomycin application of electric pulses (8 pulses, duration 100 microseconds, frequency 8 Hz with amplitude adequate to cover the whole treated lesion with electric field necessary for reversible plasma membrane permeabilization), removal of electrodes.
  The maximum duration of procedure is 90 minutes, after liver mobilization.
  Bleomycin PHC 15 e. (United States Pharmacopeia - USP): Intravenous in bolus administration of bleomycin (15 mg/m2)
Period: Overall Study
Arm/Group | Electrochemotherapy Treatment
Started | 25
Completed | 24
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Electrochemotherapy Treatment
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 15
Age, Continuous [Median (Full Range); unit: years] | 65.6 [52 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Toxicity Related to Electrochemotherapy
Description: Biochemistry, blood test and/or US
Time Frame: After operation on day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Electrochemotherapy Treatment
Number analyzed (Participants) | 24
Participants
  No adverse events | 20
  ECT-related adverse events | 0
  Non-ECT-related within 24 h | 0
  Non-ECT-related after 24 h | 4

2. Secondary Outcome: Clinical Response Evaluation According to RECIST v1.1
Description: Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI/CT:
  Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: After operation on days 1, 7, 30, 60, 90, 120
Measure: Count of Participants; unit: Participants
Arm/Group | Electrochemotherapy Treatment
Number analyzed (Participants) | 24
Participants
  complete response (CR) | 19
  partial response (PR) | 4
  stable disease (SD) | 1
  progressive disease (PD) | 0

ADVERSE EVENTS:
Time Frame: 7, 30, 60, 90, 120 days
Arm/Group | Electrochemotherapy Treatment
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 15/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Electrochemotherapy Treatment (N=24)
Clavien-Dindo Classification, Grade I (General disorders) | 11 (11)
Clavien-Dindo Classification, Grade II (Hepatobiliary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2014-11-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT02291133/Prot_SAP_ICF_000.pdf